CLINICAL TRIAL: NCT00990756
Title: A Double Blind (3rd Party Open), Randomised, Placebo Controlled, Dose Escalation Study To Investigate The Safety, Toleration, And Pharmacokinetics Of Multiple Inhaled Doses Of PF-03526299 In Healthy Male Subjects
Brief Title: A Phase 1 Study To Evaluate The Safety And Tolerability Of Different Doses Of PF-03526299 In Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: A9291003
Record Dates: First submitted 2009-10-05; First posted 2009-10-07 (Estimated); Last update posted 2010-01-22 (Estimated); Status verified 2010-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-03526299 1.396 mg (Experimental)
  Interventions: Drug: PF-03526299
- PF-03526299 4mg (Experimental)
  Interventions: Drug: PF-03526299

INTERVENTIONS:
Drug: PF-03526299 — dry powder for inhalation, 1.396 mg, BID for 14 days
  Arms: PF-03526299 1.396 mg
Drug: PF-03526299 — dry powder for inhalation, 4 mg, BID for 14 days
  Arms: PF-03526299 4mg

SUMMARY:
The purpose of this study is to investigate safety and toleration of multiple inhaled doses as well as the time course of PF-03526299 concentration in the blood following dosing by dry powder inhaler.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects and females of non-childbearing potential between the ages of 21 and 55 years.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m^2; and a total body weight >50 kg (110 lbs).
* Subjects who had a normal chest X-ray in the previous 6 months prior to Screening

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* A positive urine drug screen.
* History of regular alcohol consumption exceeding 21 drinks/week for males and 14 drinks/week for females.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Safety/toleration: Adverse events, vital signs, 12 lead ECG, blood and urine safety tests and physical examination. | 17 days

SECONDARY OUTCOMES:
Pharmacokinetic parameters: Plasma Day 1: Cmax, Tmax, AUCτau. | Day 1 - 17
Plasma Day 7: Cmax, Tmax. | 7 Days
Plasma Day 14: Cmax, Tmax, CL/F, AUCτau, t½, accumulation ratio, time to steady state. | 14 Days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9291003&StudyName=A%20Phase%201%20Study%20To%20Evaluate%20The%20Safety%20And%20Tolerability%20Of%20Different%20Doses%20Of%20PF-03526299%20In%20Healthy%20Adult%20Volunteers